CLINICAL TRIAL: NCT00005998
Title: Autologous Transplantation for Non-Hodgkin's Lymphoma and Hodgkin's Disease Using Retrovirally Marked Peripheral Blood Progenitor Cells Obtained After In Vivo Mobilization Using Hematopoietic Cytokines Plus Chemotherapy
Brief Title: Peripheral Stem Cell Transplantation With Specially Treated Stem Cells in Treating Patients With Non-Hodgkin's Lymphoma or Hodgkin's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn because study never enrolled patients
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: 1999LS080; MT1999-19 (Other: Blood and Marrow Transplantation Program); NCI-G00-1807
Record Dates: First submitted 2000-07-05; First posted 2003-10-08 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Carmustine; Cyclophosphamide; Cytarabine; Dexamethasone; Etoposide; Filgrastim; Mitoxantrone; Peripheral Blood Stem Cell Transplantation; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: carmustine
Drug: cyclophosphamide
Drug: cytarabine
Drug: dexamethasone
Drug: etoposide
Drug: filgrastim
Drug: mitoxantrone hydrochloride
Drug: retrovirus vector LN
Procedure: in vitro-treated peripheral blood stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Procedure: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Combining chemotherapy and radiation therapy with peripheral stem cell transplantation using specially treated stem cells may allow the doctor to give higher doses of chemotherapy drugs and radiation therapy and kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of peripheral stem cell transplantation using specially treated stem cells in treating patients who have non-Hodgkin's lymphoma or Hodgkin's disease.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether priming with hematopoietic cytokines and chemotherapy increases the yield of hematopoietic progenitors in peripheral blood stem cells (PBSC) in patients with non-Hodgkin's lymphoma or Hodgkin's disease undergoing autologous PBSC transplantation.
* Determine whether in vitro studies can predict the transduction efficiency of early and late engrafting hematopoietic stem cells in this patient population undergoing this treatment.
* Determine whether in vitro transduction of a graft product stable long term transduction of marrow cells in these patients after autologous transplantation.

OUTLINE: Patients receive filgrastim (G-CSF) subcutaneously (SC) twice daily on days 1-7. Peripheral blood stem cells (PBSC) are collected on days 5-7. Patients receive cyclophosphamide IV over 2 hours, mitoxantrone IV, and cytarabine IV every 12 hours for 2 doses on day 10, and dexamethasone every 12 hours for 4 doses on days 10 and 11. Patients receive G-CSF SC for the next 10-20 days. Additional PBSC are collected on days 25-28 or 29. Beginning 7 days before PBSC transplantation, patients receive cyclophosphamide IV over 2 hours on days -7 and -6 and total body irradiation (TBI) twice daily on days -4 to -1. Patients unable to tolerate TBI receive cyclophosphamide IV over 2 hours on days -6 to -3, carmustine IV over 1 hour on days -6, and etoposide IV over 1 hour every 12 hours on days -6 to -4. Retrovirally transduced PBSC are reinfused on day 0 followed by another course of G-CSF SC until hematopoietic recovery.

Patients are followed at 1, 3, 6, 9, 12, 18, and 24 months and then annually thereafter.

PROJECTED ACCRUAL: A total of 15-20 patients will be accrued for this study within 12-15 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Intermediate or high grade non-Hodgkin's lymphoma (NHL) or Hodgkin's disease (HD)

  * Chemotherapy sensitive, initial partial remission OR
  * Relapse after initial complete or partial remission
* Low grade NHL eligible provided progression following initial partial or complete remission
* Ineligible for ongoing allogeneic marrow donor transplant protocols or elected not to participate in such protocols
* No chemotherapy resistant NHL or HD NOTE: A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Performance status:

* Karnofsky 90-100%

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* AST less than 2.5 times upper limit of normal (ULN)
* Bilirubin less than 2.5 times ULN

Renal:

* Creatinine less than 2.0 mg/dL

Cardiovascular:

* Resting LVEF at least 40%
* No unstable ischemic heart disease

Pulmonary:

* Spirometry and DLCO greater than 50% predicted

Other:

* No active uncontrolled infection
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2000-01; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Weisdorf, MD, Study Chair — Masonic Cancer Center, University of Minnesota